CLINICAL TRIAL: NCT00809731
Title: A Naturalistic Observational Study to Evaluate Efficacy of 2nd-generation Antipsychotics and Remission Status for Patients With Schizophrenia / Schizoaffective Disorder
Brief Title: Observational Study to Evaluate Efficacy and Remission Status for Schizophrenia Patients Under Atypical Treatment
Acronym: QTP NIS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Robin Meng/Marketing Company Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-NTW-SER-2008/1
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia remission status by 8-item PANSS
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational Group: All commercially available 2nd-generation antipsychotic with an indication of treating schizophrenia will be prescribed by the physician according to normal practices

SUMMARY:
The objective of this study is to evaluate under routine clinical setting the efficacy and remission status from treatment of 2nd-generation antipsychotic in patients who is upon acute episode or not achieving remission under regular treatment from schizophrenia/schizoaffective disorder. This study will collect in real-life practice the severity of schizophrenia by Clinical Global Impression (CGI), also evaluate the criteria of schizophrenia remission applying 8 items of Positive and Negative Syndrome Scale (PANSS) from Andresen working group, the Montgomery and Asberg Depression Rating Scale (MADRS), and the Global Assessment of Functioning Scale (GAF). Side effect of movement disorder will be evaluated by Drug Induced Extrapyramidal Symptoms Scale (DIEPSS). Tolerability for treatment will be monitored by documenting spontaneous reports on adverse events as well as change in body weight.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute episode (first or relapse), or upon revisit and identified not achieving remission of schizophrenia or schizoaffective disorder (according to remission criteria of schizophrenia)
* Male or female aged between 18 and 65 years
* Patients recruited from both in-patient and out-patient clinics
* Patients who are cooperative, by judgment from investigators, and the use of oral antipsychotic considered adequate

Exclusion Criteria:

* Pregnancy or lactation
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Known intolerance, lack of response, or contraindication to prescribed atypical antipsychotic, as judged by the investigator
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before enrolment and patients prescribed with clozapine within 3 months prior to enrolment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute episode (first or relapse), or upon revisit and identified not achieving remission of schizophrenia or schizoaffective disorder (according to remission criteria of schizophrenia)
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
CGI-Severity of illness (CGI-SI) | Visit 1(Day 0), 2(Day 3), 3(Week 1), 4(Week 2), 5(Week 4)

SECONDARY OUTCOMES:
CGI-Degree of change (CGI-DC) | Visit 2(Day 3), 3(Week 1), 4(Week 2), 5(Week 4)
MADRS, GAF, DIEPSS | Visit 1(Day 0), 2(Day 3), 3(Week 1), 4(Week 2), 5(Week 4)
Remission status | Visit 1(Day 0), 5(Week 4)

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Hwa Chou, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (17):
- Taiwan (17):
  - Research Site, Changhua
  - Research Site, Changhua-Lugang
  - Research Site, Chiayi City
  - Research Site, Kaohsiung-Niosong
  - Research Site, Kaohsiung-Sanmin
  - Research Site, Kaohsiung-Yanchao
  - Research Site, Keelung
  - Research Site, Miaoli
  - Research Site, Miaoli-Toufen
  - Research Site, Taichung-Beitun
  - Research Site, Taichung-Shalu
  - Research Site, Taipei-Banciao
  - Research Site, Taipei-Datong
  - Research Site, Taipei-Shilin
  - Research Site, Taipei-Shipai
  - Research Site, Taipei-Xindian
  - Research Site, Taoyuan District